CLINICAL TRIAL: NCT05041309
Title: Long-term Follow-up Study for Participants of Kite-Sponsored Interventional Studies Treated With Gene-Modified Cells
Status: Enrolling by invitation | Type: Observational
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Other Study IDs: KT-US-982-5968; 2020-005843-21 (EudraCT Number); MOH_2022-08-21_010606 (Registry Identifier: Israel Clinical Research Site); 2023-507041-28 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2021-08-27; First posted 2021-09-13 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Solid and Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — axicabtagene ciloleucel; brexucabtagene autoleucel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh or archival tumor samples, bone marrow biopsy and/or aspirate and blood draws
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Axicabtagene Ciloleucel (KTE-C19): All participants who previously received axicabtagene ciloleucel (KTE-C19) in the parent study will be enrolled in this cohort for long-term follow-up.
  Interventions: Biological: Axicabtagene Ciloleucel
- Brexucabtagene Autoleucel (KTE-X19): All participants who previously received brexucabtagene autoleucel (KTE-X19) in the parent study will be enrolled in this cohort for long-term follow-up.
  Interventions: Biological: Brexucabtagene Autoleucel
- Anitocabtagene autleucel: All participants who previously received anitocabtagene autleucel in the parent study will be enrolled in this cohort for long-term follow-up.
  Interventions: Biological: Anitocabtagene autleucel
- KITE-753: All participants who previously received KITE-753 in the parent study will be enrolled in this cohort for long-term follow-up.
  Interventions: Biological: KITE-753
- KITE-197: All participants who previously received KITE-197 in the parent study will be enrolled in this cohort for long-term follow-up.
  Interventions: Biological: KITE-197
- KITE-363: All participants who previously received KITE-363 in the parent study will be enrolled in this cohort for long-term follow-up.
  Interventions: Biological: KITE-363

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — No investigational product will be administered
  Other Names: Yescarta®
  Groups: Axicabtagene Ciloleucel (KTE-C19)
Biological: Brexucabtagene Autoleucel — No investigational product will be administered
  Other Names: Tecartus™
  Groups: Brexucabtagene Autoleucel (KTE-X19)
Biological: Anitocabtagene autleucel — No investigational product will be administered
  Other Names: CART-ddBCMA
  Groups: Anitocabtagene autleucel
Biological: KITE-753 — No investigational product will be administered
  Groups: KITE-753
Biological: KITE-197 — No investigational product will be administered
  Groups: KITE-197
Biological: KITE-363 — No investigational product will be administered
  Groups: KITE-363

SUMMARY:
The goal of this clinical study is to learn more about the long-term safety, effectiveness and prolonged action of Kite study drugs, axicabtagene ciloleucel, brexucabtagene autoleucel, KITE-363, KITE-753, KITE-197, and anitocabtagene autoleucel in participants of Kite-sponsored interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* The individual must have received an infusion of gene-modified cells in a completed Kite-sponsored parent study, has not withdrawn full consent, and has discontinued or completed the post-treatment follow-up period in the parent study, as applicable
* The individual must understand and voluntarily sign an Informed Consent Form (ICF) or an Informed Assent Form prior to any study-related assessments or procedures being conducted
* In the investigator's judgment, the individual is willing and able to complete the protocol-required follow-up schedule and comply with the study requirements for participation

Exclusion Criteria: none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants who received an infusion of gene-modified cells and have not died, withdrawn consent, been withdrawn by the investigator, or been lost to follow-up at the time of transition from the completed parent study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Late-onset Targeted Adverse Events (AEs) | Up to 15 years
  Targeted AEs include late-onset targeted AEs suspected to be possibly related to gene-modified cells include neurologic disorders, autoimmune disorders, hematologic disorders, serious infections, and new malignancies.
Percentage of Participants Experiencing Late-onset Targeted Serious Adverse Events (SAEs) | Up to 15 years
  Targeted SAEs include late-onset targeted SAEs suspected to be possibly related to gene-modified cells include neurologic disorders, autoimmune disorders, hematologic disorders, serious infections, and new malignancies.
Height of Pediatric and Adolescent Participants | Up to 15 years
Weight of Pediatric and Adolescent Participants | Up to 15 years
Sexual Maturation of Pediatric and Adolescent Participants Assessed by Tanner Pubertal Stage Scale Score | Up to 15 years
  The Tanner Pubertal Stage Scale is a measure of pubertal development (sexual maturation) in children and adolescents with components described for each sex, rated separately on a scale of stage one to stage five, with 1 for preadolescent and 5 for mature/adult.

SECONDARY OUTCOMES:
Time to Subsequent Anticancer Therapies | Up to 15 years
  Time to subsequent anticancer therapies will be assessed only per regulatory request or sponsor needs.
Survival Status Assessment | Up to 15 years
  Survival status will be assessed as the length of time from the participant's first dose date of study drug to death during the study due to any cause or last date of being alive during the study. Survival status will be assessed only per regulatory request or sponsor needs.
Percentage of Participants With Cause of Death | Up to 15 years
Overall Rate of Replication-competent Retrovirus/Replication-competent Lentivirus (RCR/RCL) | Up to 15 years
Percentage of Participants With Vector Integration Site(s) for Replication-competent Retrovirus/Replication-competent Lentivirus (RCR/RCL) or Insertional Mutagenesis for Confirmed Events Related to the Cell Therapy Product | Up to 15 years
Percentage of Participants With Status of Primary Malignant Disease | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (87):
- United States (47):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Sylvester Comprehensive Cancer Centre, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Ann& Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago Medical Center Clinical Laboratories, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Cancer Center Westwood, Westwood, Kansas
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center Institute, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ichann School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Mayo Clinic, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - DUHS-Duke Blood Cancer Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Sarah Cannon-Methodist Healthcare System - San Antonio, San Antonio, Texas
  - Intermountain LDS Hospita;/Blood and Marrow Transplant/ Acute Leukemia Program, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Medizinische Universitat Innsbruck, Innere Medizin V - Hamatologie und Onkologie, Innsbruck, Austria
- UZ Leuven, Leuven, Belgium
- Canada (6):
  - McGill University Health Center, Montreal
  - The Ottawa Hospital - General Campus, Ottawa
  - Hôpital de l'Enfant-Jésus, Québec
  - The hospital for sick children, Toronto
  - Princess Margaret Cancer Center - University Health Network, Toronto
  - Vancouver General Hospital, Vancouver
- France (6):
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Hospital Saint Eloi, Montpellier
  - Hopital Saint-Louis, Paris
  - CHU Bordeaux, Hopital Haut-Leveque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Hôpital Pontchaillou - CHU de Rennes, Rennes
- Germany (6):
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universittsklinikum Heidelberg, Heidelberg
  - Johannes Gutenberg University Hospital-University Mainz, Mainz
  - LMU Klinikum der Universitat Munchen,Med. Klinik und Poliklinik III, München
  - Universitatsklinikum Wurzburg, Med. Klinik und Poliklinik II, Zentrum lnnere Medizin, Würzburg
- Tel Aviv Souraski Medical Center, Tel Aviv, Israel
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy
- Japan (5):
  - Kyushu University Hospital, Fukuoka
  - Kyoto University Hospital, Kyoto
  - Okayama University Hospital, Okayama
  - Hokkaido University Hospital, Sapporo Hokkaido
  - National Cancer Center Hospital, Tokyo
- Netherlands (5):
  - Amsterdam Universitair Medische Centra (UMC), Amsterdam
  - University Medical Centre Groningen, Groningen
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus University Medical Centre (MC), Rotterdam
  - UMC Utrecht, Utrecht
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catalia d'Oncologia L'Hospitalet, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
- Istituto Oncologico Della Svizzera Italiana (IOSI), Bellinzona, Switzerland
- United Kingdom (2):
  - King's College Hospital, London
  - The Royal Marsden NHS Foundation Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KT-US-982-5968